CLINICAL TRIAL: NCT04952701
Title: Evaluating the Success of Habitual Multifocal Wearers When Refit With a New Lens Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-119
Record Dates: First submitted 2021-06-28; First posted 2021-07-07 (Actual); Results first posted 2022-04-26 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control Lens (Active Comparator): All subjects will wear control lenses for two weeks and then will wear Test lenses for two weeks.
  Interventions: Device: Control lenses; Device: Test lenses
- Test Lens (Experimental): After wearing control lenses for two weeks, all subjects will wear test lenses for two weeks.
  Interventions: Device: Control lenses; Device: Test lenses

INTERVENTIONS:
Device: Control lenses — Control Multifocal lenses
Device: Test lenses — Test Multifocal lenses

SUMMARY:
The objective of the study was to adapt existing multifocal soft lens wearers to a CONTROL lens for 2 weeks and then evaluate the success of switching them to the TEST lens, with a review after 2 weeks.

DETAILED DESCRIPTION:
This was a prospective, crossover, bilateral daily wear, and subject masked dispensing study. The habitual contact lenses were not optimized. There was no randomization of the study lenses, participants wore the control lenses for the first wear period and the test for the second wear period. Participants wore each study lens for 3-7 days and then attend a prescription optimization visit. After this optimization visit, they wore each study lens for a 2-week period. During the 2-week wear period, participants recorded their subjective lens-wear experience remotely.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 42 years of age and has full legal capacity to volunteer;
2. Has read and signed an information consent letter;
3. Self reports having a full eye examination in the previous two years;
4. Anticipates being able to wear the study lenses for at least 8 hours a day, 5 days a week;
5. Is willing and able to follow instructions and maintain the appointment schedule;
6. Habitually wears multifocal soft contact lenses, for the past 3 months minimum;
7. Has refractive astigmatism no higher than -0.75DC;
8. Is presbyopic and requires a reading addition of at least +0.75D and no more than

   +2.50D;
9. Can be fit and achieve binocular distance vision of at least 20/30 Snellen (or +0.20 logMAR) which participants also deem to be 'acceptable', with the available study lens parameters (powers +4.00 to -6.00DS)

Exclusion Criteria:

1. Is participating in any concurrent clinical or research study;
2. Has any known active* ocular disease and/or infection that contraindicates contact lens wear;
3. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
4. Is using any systemic or topical medications that in the opinion of the investigator may affect contact lens wear or a study outcome variable;
5. Has known sensitivity to the diagnostic sodium fluorescein used in the study;
6. Self-reports as pregnant, lactating or planning a pregnancy at the time of enrolment;
7. Has undergone refractive error surgery or intraocular surgery.

Min Age: 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, Study Director — University of Waterloo
Locations (5):
- United States (5):
  - Coan EyeCare, Ocoee, Florida
  - Kannarr Eye care, Pittsburg, Kansas
  - Sacco Eye Group PLLC, Vestal, New York
  - ProCare Vision Center, Granville, Ohio
  - Nittany Eye Associates, College, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: All subjects wore control lenses for two weeks and then wore Test lenses for two weeks.
  Control lenses: Control Multifocal lenses
  Test lenses: Test Multifocal lenses
Period: Control Lens
Arm/Group | Overall Study
Started | 63
Completed | 59
Not Completed | 4
Not completed — Physician Decision | 4
Period: Test Lens
Arm/Group | Overall Study
Started | 59
Completed | 58
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: All subjects wore control lenses for two weeks and then test lenses for two weeks.
Arm/Group | Overall Study
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 63
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 63

OUTCOME MEASURES:

1. Primary Outcome: Comfort on Insertion
Description: Subjective ratings of comfort on insertion using a 0-10 scale, in 0.5 steps (0=- painful, 10- Can't feel the lenses).
Time Frame: Day 1 after Lens Dispense Visit
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control Lens: All subjects wore control lenses for two weeks.
  Control lenses: Control Multifocal lenses
- Test Lens: All subjects wore test lenses for two weeks.
  Test lenses: Test Multifocal lenses
Arm/Group | Control Lens | Test Lens
Number analyzed (Participants) | 58 | 58
units on a scale | 9.2 (1.1) | 9.2 (1.0)

ADVERSE EVENTS:
Time Frame: From dispense up to 2 weeks on each study lens, a total of 4 weeks.
Groups:
- Control Lens: All subjects wore control lenses for two weeks and then wore Test lenses for two weeks.
  Control lenses: Control Multifocal lenses
- Test Lens: After wearing control lenses for two weeks, all subjects wore test lenses for two weeks.
  Test lenses: Test Multifocal lenses
Arm/Group | Control Lens | Test Lens
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/63
Other Adverse Events (participants affected / at risk) | 2/63 | 2/63
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Lens (N=63) | Test Lens (N=63)
Light Sensitivity (Eye disorders) | 2 (2) | 0
Eye Irritation and Discomfort (Eye disorders) | 0 | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/01/NCT04952701/Prot_SAP_000.pdf